CLINICAL TRIAL: NCT04664894
Title: New Drugs And New Concerns: Gaining Insight Through Pharmacovigilance Of Direct Acting Anti-Viral's In Chronic HCV Patients
Brief Title: Direct Acting Anti-Viral's In Chronic HCV Patients
Status: Completed | Type: Observational
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GTZ-NLRF-001
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Safety Issues
Keywords: adverse events; chronic hepatitis; direct acting antivirals
MeSH Terms: conditions — Hepatitis, Chronic | interventions — Sofosbuvir; daclatasvir; Ribavirin; velpatasvir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sofosbuvir — the occurrence of AEs (AE) and their severity among chronic HCV patients has assessed in patinets receiving different combinations of DAAs in Pakistani Population
  Other Names: Daclatasvir; Ribavirin; Velpatasvir

SUMMARY:
The objective of the study is to determine the safety of DAA's among chronic HCV patients. The outcomes of the study are; To determine the frequency of adverse events while receiving DAAs with or without RBV and/or Pegylated Interferon To calculate the percentage of patients with severity of medical event as per Karch and Lasagna classification To determine the percentage of patient having serious adverse event as per ICH Classification

DETAILED DESCRIPTION:
The cross sectional survey data will be collected on a pre-defined questionnaire from Gastroenterologist and Hepatologist. The questionnaire will provide us information on demographics, relevant patient history, concomitant medication, ongoing treatment plan recommended for chronic HCV and adverse event details.

The questions related to Pharmacovigilance and safety assessment includes the International Nonproprietary Names (INN) unless it is prescribed brand of Getz Pharma. All adverse events associated with the prescribed treatment will be recorded. Data on outcome assessment will be based on action taken due to AE and other reported details. Seriousness of adverse event will also be recorded as per the ICH classification and severity of medical event will be assessed as per Karch and Lasagna classification.

All the information will be recorded by the healthcare professionals on the questionnaire during direct interaction with the patients.

Patients' written authorization to use and/or disclose the patient's personal and/or health data will be obtained. However, patient data secrecy will follow ICH GCP requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or Female patient
3. Age of patient ≥18 years
4. Patients already diagnosed with HCV and on DAAs therapy.

Exclusion Criteria:

1. Written informed consent
2. Male or Female patient
3. Age of patient ≥18 years
4. Patients already diagnosed with HCV and on DAAs therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C on DAAs therapy were included. The primary inclusion criteria was both gender with age >18years and written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events while receiving DAAs with or without RBV and/or Pegylated Interferon | 12 months
  Frequency of adverse events while receiving DAAs with or without RBV and/or Pegylated Interferon

SECONDARY OUTCOMES:
Percentage of patients reported severity of medical event as per Karch and Lasagna classification | 12 months
  Percentage of patients reported severity of medical event as per Karch and Lasagna classification

OTHER OUTCOMES:
Percentage of patient having serious adverse event as per ICH Classification | 12 months
  Percentage of patient having serious adverse event as per ICH Classification

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Center Faisalabad, Faisalabad, Punjab Province, Pakistan